CLINICAL TRIAL: NCT04918875
Title: Oxygen Requirements and Approaches to Respiratory Support in Patients With COVID-19 in LMICs: A WHO Study
Brief Title: Oxygen Requirements and Use in Patients With COVID-19 in LMICs
Acronym: O2CoV2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pryanka Relan (Other)
Responsible Party: Sponsor-Investigator, Pryanka Relan, Technical officer, World Health Organization
Organization: World Health Organization (Other)
Other Study IDs: CERC.0040
Record Dates: First submitted 2021-05-31; First posted 2021-06-09 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Covid19; COVID-19 Pneumonia
Keywords: oxygen; covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients 12 years of age or older with suspected or confirmed COVID-19, deemed to require oxygen.

SUMMARY:
This observational cohort study will enroll patients in LMICs with suspected or confirmed COVID-19 on oxygen or deemed to require oxygen therapy based on objective criteria. Demographics and risk factor information will be collected from participants. Participants will be followed for 7 days or until outcome (hospital discharge or death). Facility level metrics on oxygen availability will also be collected at the beginning of site enrolment.

DETAILED DESCRIPTION:
The COVID-19 pandemic has highlighted, more than ever, the acute need for scale up of oxygen therapy. WHO has provided an inventory tool to quantify facility-level provision of infrastructure to deliver oxygen therapy. However, data on the use of oxygen therapy at the patient-level remains lacking. This observational cohort study will enroll patients in LMICs with suspected or confirmed COVID-19 on oxygen or deemed to require oxygen therapy based on objective criteria. Demographics and risk factor information will be collected from participants. Participants will be followed for 7 days or until outcome (hospital discharge or death). Facility level metrics on oxygen availability will also be collected at the beginning of site enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected SARS-CoV-2 infection as determined by treating clinical provider, or confirmed SARS-CoV-2 infection confirmed virologically in the lab by RT-PCR via nasopharyngeal or oropharyngeal sample or by SARS-CoV-2 Ag-RDTs that meet the minimum performance requirements of ≥80% sensitivity and ≥97% specificity compared to a NAAT reference assay.
2. Receiving supplemental oxygen or showing clinical evidence of need for supplemental respiratory support as reflected in a respiratory rate ≥30 breaths per minute or an SpO2 ≤ 90%, SpO2 < 94 % if any emergency signs are present
3. Admitted to health care facility

Exclusion Criteria:

1. Is not receiving oxygen or does not have clinical criteria for oxygen treatment specified above oxygen therapy
2. Does not have suspected or confirmed COVID-19 (as per criteria above)
3. Patient younger than 12 years of age
4. Lack of commitment to full supportive care

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who access emergency unit/department (if available) or anywhere acutely ill patients are first assessed.
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients receiving oxygen via each of various delivery devices. | Over first 7 days of hospitalization
  Oxygen delivery devices analysed: nasal cannulae, face mask, Venturi, NRB, HFNO, CPAP, NIV, IMV
Proportion of patients progressing to invasive mechanical ventilation | Over first 7 days of hospitalization
  If available at facility
Total oxygen requirements in patients receiving oxygen via each of various delivery devices. | Over first 7 days of hospitalization
  Daily oxygen use measured in liters.
  For nasal cannula, facemask, and non-rebreather FiO2 is assumed to be 1.0 and flow rates are adjustable in liters per minute. Liter per day consumption of O2 = device flow rate L/minute x 60 minutes/hr x 24 hr/day For high flow nasal cannula FiO2 is adjustable (defaulted to 1.0) and flow rate is adjustable in liters per minute.
  Liter per day consumption of O2 = device flow rate L/minute x 60 minutes/hr x 24 hr/day; flow rate in LPM = device flow rate x (FiO2 - 0.21)/0.79 For ventilator, CPAP, BIPAP/NIPPV FiO2 is adjustable (defaulted to 1.0) and flow rate is adjustable in liters per minute and dependent on multiple factors. Liter per day consumption of O2 = device O2 consumption rate L/minute x 60 minutes/hr x 24 hr/day Device O2 consumption rate in LPM = (Minute ventilation + (bias flow x RR x expiratory time/60) + leak) x (FiO2 - 0.21)/0.79

SECONDARY OUTCOMES:
Demographics and outcomes at hospital discharge of cohort of hospitalized patients | Until patient discharge from hospital or death, censored at 30 days.
  Baseline characteristics, daily parameters over 7 days, hospital outcomes
Quantification of total oxygen supply at each facility | One time at beginning of enrolment
  Description of oxygen source, distribution and biomedical equipment at facility level and estimated oxygen capacity at the facility level

CONTACTS AND LOCATIONS:
Overall Officials: WHO, Study Director — World Health Organization
Locations (1):
- World Health Organization, Geneva, Other, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Relan P, Rylance J, Arabi YM, Convocar P, Rolland M, Diaz JV; O2CoV2 investigators. Medical oxygen and respiratory support requirements for patients hospitalised with COVID-19 in 23 low-income and middle-income countries: a prospective, observational cohort study. Lancet Glob Health. 2026 Feb;14(2):e233-e241. doi: 10.1016/S2214-109X(25)00480-2. PMID 41519152
- [Derived] Relan P, Murthy S, Marshall JC, Annane D, Chevret S, Arabi YM, Waweru-Siika W, Dominguez Rodriguez S, Convocar P, Diaz J; World Health Organization Respiratory Support Research Group; World Health Organization O2CoV2 International Study Steering Committee. WHO O2CoV2: oxygen requirements and respiratory support in patients with COVID-19 in low-and-middle income countries-protocol for a multicountry, prospective, observational cohort study. BMJ Open. 2023 Aug 17;13(8):e071346. doi: 10.1136/bmjopen-2022-071346. PMID 37591648